CLINICAL TRIAL: NCT04550936
Title: Patterns of Real-World Isavuconazole Use, Effectiveness, Safety, and Healthcare Resource Utilization-a Retrospective Chart Review Study of Patients With Mucormycosis or Invasive Aspergillosis (PRISMA)
Brief Title: A Study to Understand How the Use of Paxlovid Affected the Healthcare Use in People With Pre-existing Conditions.
Acronym: PRISMA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3791008; NCT04550936 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Invasive Aspergillosis; Mucormycosis
MeSH Terms: conditions — Mucormycosis | interventions — isavuconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Isavuconazole — antifungal agent
  Other Names: Cresemba

SUMMARY:
This is a non-interventional medical chart review study aiming to examine the effectiveness, safety, and treatment patterns of isavuconazole in 5 European countries (France, Germany, Italy, Spain, and United Kingdom). Eligible patients are adults who have been treated with isavuconazole in routine practice at participating sites since 15 October, 2015 or since the date of launch in the country if it is after 15 October, 2015 until 30 June, 2019. As this is an observational study, patients will be treated based on the standard of care at the discretion of their physician. No drugs will be supplied for this study and patients will receive treatment through standard local practice.

DETAILED DESCRIPTION:
This observational study will include approximately 600 patients diagnosed with invasive aspergillosis or mucormycosis who received treatment with at least one dose of isavuconazole in the hospital setting.

Patients will be recruited in approximately 20 sites across 5 countries in Europe. Patients will be followed from isavuconazole initiation (index event) until six-months post-index treatment discontinuation, death, loss to follow-up, or 31 December, 2019, whichever occurs first.

De-identified data on patient demographics, disease characteristics, treatment effectiveness, safety outcomes, isavuconazole treatment patterns, and HCRU will be collected from patient medical records and entered into an electronic data capture (EDC) system by site staff. Follow-up data will include details of treatment over time and clinical, radiological, mycological, and healthcare resource utilization outcomes. As this study is retrospective, information pertaining to patient care will already be documented in patient medical records at the time of chart abstraction.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patient must be aged ≥ 18 years at the time of isavuconazole initiation
2. Patient must have a record of a diagnosis of invasive aspergillosis or mucormycosis in their medical record at the time isavuconazole was initiated (regardless of whether this diagnosis is suspected or confirmed )
3. Patient must have received at least one dose of isavuconazole during the eligibility period (October 15, 2015, to June 30, 2019)

Exclusion Criteria:

1. Patients who did not receive at least one dose of isavuconazole for treatment of invasive aspergillosis or mucormycosis within the eligibility period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who received isavuconazole for the treatment of invasive aspergillosis or mucormycosis in the hospital setting in five European countries (France, Germany, Italy, Spain, and the United Kingdom).
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- France (3):
  - CHU de Limoges, Limoges
  - Paris University, Paris
  - Institut de Cancérologie, Strasbourg
- Germany (4):
  - University Hospital of Cologne, Cologne
  - Universitätsklinik Frankfurt, Frankfurt
  - Klinikum rechts der Isar Technische Universität München, Munich
  - Comprehensive Cancer Center Ulm (CCCU), Ulm
- Azienda Ospedaliero Universitaria Città della Salute e della Scienza di Torino, Turin, Piedmont, Italy
- Spain (5):
  - Vall d'Hebron University Hospital, Barcelona
  - Fundació Clínic Per A La Recerca Biomèdica, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - University Hospital Miguel Servet, Zaragoza
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - King'S College Hospital Nhs Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Neofytos D, Pagliuca A, Houghton K, Broughton E, de Figueiredo Valente MLN, Jiang L, Enoch DA, Gruener B, Herbrecht R, Lahmer T, Lortholary O, Melenotte C, De Rosa FG, Garcia-Vidal C, Jimenez M, Fernandez M, Cornely O. Effectiveness, Safety, and Patterns of Real-World Isavuconazole Use in Europe (2015-2019). Infect Dis Ther. 2024 Dec;13(12):2527-2543. doi: 10.1007/s40121-024-01064-4. Epub 2024 Oct 24. PMID 39443403
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3791008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from the medical records of participants with invasive aspergillosis or mucormycosis who initiated isavuconazole treatment during the index period of 15 October 2015 until 30 June 2019 were included in this study.
Pre-assignment Details: Retrospective data was extracted and evaluated from study start date and until study completion (approximately 34 months) of this retrospective observational study. Participants were followed from index date until 6 months post-index treatment discontinuation, death, loss to follow-up, whichever occurs first.
Groups:
- Invasive Aspergillosis: Participants with aspergillosis who received isavuconazole treatment in between 15-Oct-2015 to 30-Jun-2019 under routine clinical practice and whose data were observed in the study, were included in this reporting group.
- Mucormycosis: Participants with mucormycosis who received isavuconazole treatment in between 15-Oct-2015 to 30-Jun-2019 under routine clinical practice and whose data were observed in the study, were included in this reporting group.
Period: Overall Study
Arm/Group | Invasive Aspergillosis | Mucormycosis
Started | 201 | 17
Completed | 201 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Invasive Aspergillosis | Mucormycosis | Total
Number analyzed (Participants) | 201 | 17 | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (15.6) | 66.5 (12.8) | 56.8 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 9 | 74
  Male | 136 | 8 | 144
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at Week 6
Description: Clinical response was evaluated according to the following mutually exclusive modalities: Clinical success, clinical failure and unknown. Clinical success: resolution or partial resolution of all attributable clinical symptoms and physical findings. Clinical failure: no resolution of any attributable clinical symptoms and physical findings and/or worsening. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any clinical response at Week 6 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: Week 6 post index date (retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 173 | 14
  Clinical success | 27 | 3
  Clinical failure | 1 | 0

2. Primary Outcome: Number of Participants With Clinical Response at Week 12
Description: Clinical response was evaluated according to the following mutually exclusive modalities: Clinical success, clinical failure and unknown. Clinical success: resolution or partial resolution of all attributable clinical symptoms and physical findings. Clinical failure: no resolution of any attributable clinical symptoms and physical findings and/or worsening. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any clinical response at Week 12 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: Week 12 post index date (retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 185 | 15
  Clinical success | 16 | 2
  Clinical failure | 0 | 0

3. Primary Outcome: Number of Participants With Clinical Response at Week 24
Description: Clinical response was evaluated according to the following mutually exclusive modalities: Clinical success, clinical failure and unknown. Clinical success: resolution or partial resolution of all attributable clinical symptoms and physical findings. Clinical failure: no resolution of any attributable clinical symptoms and physical findings and/or worsening. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any clinical response at Week 24 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: Week 24 post index date (retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 193 | 17
  Clinical success | 8 | 0
  Clinical failure | 0 | 0

4. Primary Outcome: Number of Participants With Radiological Response at Week 6
Description: Radiological response was evaluated according to the following mutually exclusive modalities: Radiological success, radiological failure and unknown. Radiological success: greater than or equal to (>=) 50 percent (%) improvement from initial assessment, or improvement of at least 25% from the initial assessment for the follow-up at 6 weeks or if end of treatment occurred before this time. Radiological failure: Failure to meet success criteria. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any radiological response at Week 6 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: Week 6 post index date or end of treatment, which ever occurred earlier (retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 188 | 14
  Radiological success | 11 | 3
  Radiological failure | 2 | 0

5. Primary Outcome: Number of Participants With Radiological Response at Week 12
Description: Radiological response was evaluated according to the following mutually exclusive modalities: Radiological success, radiological failure and unknown. Radiological success: >= 50% improvement from initial assessment, or improvement of at least 25% from the initial assessment for the follow-up at 12 weeks or if end of treatment occurred before this time. Radiological failure: Failure to meet success criteria. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any radiological response at Week 12 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: Week 12 post index date or end of treatment, which ever occurred earlier (retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 190 | 16
  Radiological success | 9 | 1
  Radiological failure | 2 | 0

6. Primary Outcome: Number of Participants With Radiological Response at Week 24
Description: Radiological response was evaluated according to the following mutually exclusive modalities: Radiological success, radiological failure and unknown. Radiological success: >= 50% improvement from initial assessment, or improvement of at least 25% from the initial assessment for the follow-up at 24 weeks or if end of treatment occurred before this time. Radiological failure: Failure to meet success criteria. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any radiological response at Week 24 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: Week 24 post index date or end of treatment, which ever occurred earlier (retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 195 | 16
  Radiological success | 4 | 0
  Radiological failure | 2 | 1

7. Primary Outcome: Number of Participants With Mycological Response at Week 6
Description: Mycological response was evaluated according to the following mutually exclusive modalities: Mycological success, mycological failure and unknown. Mycological success: eradication or presumed eradication of the original causative organism cultured. Mycological failure: persistence or presumed persistence. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any mycological response at Week 6 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 190 | 17
  Mycological Success: Presumed eradication | 7 | 0
  Mycological Success: Eradication | 4 | 0
  Mycological Failure | 0 | 0

8. Primary Outcome: Number of Participants With Mycological Response at Week 12
Description: Mycological response was evaluated according to the following mutually exclusive modalities: Mycological success, mycological failure and unknown. Mycological success: eradication or presumed eradication of the original causative organism cultured. Mycological failure: persistence or presumed persistence. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any mycological response at Week 12 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 2
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 195 | 17
  Mycological Success: Presumed eradication | 3 | 0
  Mycological Success: Eradication | 3 | 0
  Mycological Failure | 0 | 0

9. Primary Outcome: Number of Participants With Mycological Response at Week 24
Description: Mycological response was evaluated according to the following mutually exclusive modalities: Mycological success, mycological failure and unknown. Mycological success: eradication or presumed eradication of the original causative organism cultured. Mycological failure: persistence or presumed persistence. Unknown: if there was not enough documentation to make the classification success or failure. Number of participants with any mycological response at Week 24 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Unknown | 198 | 17
  Mycological Success: Presumed eradication | 1 | 0
  Mycological Success: Eradication | 0 | 0
  Mycological Failure | 2 | 0

10. Primary Outcome: All-Cause Mortality at Week 6
Description: Number of participants who died due to any cause at Week 6 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 48 | 1

11. Primary Outcome: All-Cause Mortality at Week 12
Description: Number of participants who died due to any cause at Week 12 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 2
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 74 | 2

12. Primary Outcome: All-Cause Mortality at Week 24
Description: Number of participants who died due to any cause at Week 24 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 3
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 93 | 5

13. Primary Outcome: Number of Participants With Adverse Event at Week 6
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Number of participants with any adverse event based on the medical records at Week 6 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 33 | 2

14. Primary Outcome: Number of Participants With Adverse Event at Week 12
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Number of participants with any adverse event based on the medical records at Week 12 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 2
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 38 | 3

15. Primary Outcome: Number of Participants With Adverse Event at Week 24
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Number of participants with any adverse event based on the medical records at Week 24 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 3
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 42 | 3

16. Primary Outcome: Number of Participants With Serious Adverse Event at Week 6
Description: Serious adverse event = any untoward medical occurrence at any dose that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, or resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect. Number of participants with any serious adverse event based on the medical records at Week 6 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 26 | 2

17. Primary Outcome: Number of Participants With Serious Adverse Event at Week 12
Description: Serious adverse event = any untoward medical occurrence at any dose that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, or resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect. Number of participants with any serious adverse event based on the medical records at Week 12 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 2
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 30 | 3

18. Primary Outcome: Number of Participants With Serious Adverse Event at Week 24
Description: Serious adverse event = any untoward medical occurrence at any dose that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, or resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect. Number of participants with any serious adverse event based on the medical records at Week 24 post index date were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 3
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 34 | 3

19. Secondary Outcome: Number of Participants According to Method of Administration
Description: Number of participants according to method of drug administration: infusion, oral and unknown were reported in this outcome measure.
Time Frame: At index date (date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019); retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Infusion | 105 | 8
  Oral | 92 | 9
  Unknown | 4 | 0

20. Secondary Outcome: Number of Participants According to Dosage of Isavuconazole Administration
Description: Number of participants according to dosage of drug administration: 200 milligram (mg), other and unknown were reported in this outcome measure.
Time Frame: as for outcome 19
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  200 mg | 186 | 17
  Other | 10 | 0
  Unknown | 5 | 0

21. Secondary Outcome: Number of Participants With Therapeutic Drug Monitoring (TDM)
Description: Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: From index date until 6 months after post-index treatment discontinuation, death, or loss to follow-up, whichever occurred first (retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 33 | 4

22. Secondary Outcome: Number of Participants With Isavuconazole Treatment Modification
Description: Treatment modification was defined as change in dose or dosing schedule of participants who received isavuconazole. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 24 | 2

23. Secondary Outcome: Number of Participants With Types of Isavuconazole Treatment Modification
Description: Number of participants with type of treatment modifications required during the index period were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 24 | 2
Participants
  Frequency decrease | 15 | 0
  Other | 14 | 1
  Change from infusion to oral capsule | 13 | 1
  Dose increase | 11 | 0
  Dose decrease | 6 | 1
  Change from oral capsule to infusion | 4 | 0
  Frequency increase | 4 | 0

24. Secondary Outcome: Duration Between Isavuconazole Treatment and Treatment Modification
Description: Duration between Isavuconazole treatment and treatment modification was defined as the date of first modification minus the date of isavuconazole treatment initiation. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 23 | 2
Days | 38.6 (59.4) | 21.5 (27.6)

25. Secondary Outcome: Percentage of Participants Who Discontinued Isavuconazole Treatment
Description: Percentage of participants who discontinued Isavuconazole treatment were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Percentage of Participants | 93.0 | 94.1

26. Secondary Outcome: Duration of Isavuconazole Treatment
Description: Duration between Isavuconazole treatment was defined as the date of discontinuation minus the date of isavuconazole treatment initiation. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 187 | 16
Days | 74.4 (121.7) | 115.6 (97.5)

27. Secondary Outcome: Number of Participants With Reasons for Isavuconazole Treatment Discontinuation
Description: Number of participants with reasons for Isavuconazole treatment discontinuation were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 187 | 16
Participants
  Death (unrelated to therapy) | 75 | 2
  Participant completed planned course of treatment | 40 | 8
  Treatment success (resolution of invasive fungal infection) | 33 | 1
  Other | 17 | 1
  Lack of response to treatment | 12 | 1
  Unknown | 9 | 1
  Adverse event | 7 | 2
  Participant decision (unrelated to AEs) | 3 | 0
  Drug-drug interaction | 3 | 0
  Therapeutic drug monitoring | 1 | 0

28. Secondary Outcome: Number of Participants Who Switched to New Antifungal
Description: Number of participants who switched to new antifungal therapy after discontinuation of Isavuconazole were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 34 | 2

29. Secondary Outcome: Number of Participants With Type of New Antifungal Therapy
Description: Number of participants according to new antifungal therapy after end of isavuconazole treatment were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 34 | 2
Participants
  Posaconazole | 12 | 1
  Liposomal amphotericin B | 10 | 1
  Voriconazole | 6 | 0
  Caspofungin | 1 | 0
  Other | 5 | 0

30. Secondary Outcome: Number of Participants With Isavuconazole Administered as Part of Combination Therapy
Description: Number of participants with index treatment administered as part of antifungal combination therapy were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019. one participant could have received more than one treatment
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 254 | 44
Participants | 53 | 27

31. Secondary Outcome: Number of Participants Who Received Other Concomitant Treatments
Description: Concomitant treatments included: Antibiotic agent, corticosteroid agent, chemotherapy, immunosuppressant agent, other and unknown were reported in this outcome measure. One participant could have more than one treatment. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 254 | 44
Participants
  Antibiotic agent | 109 | 16
  Corticosteroid agent | 17 | 2
  Chemotherapy | 7 | 2
  Immunosuppressant agent | 3 | 1
  Other | 5 | 3
  Unknown | 2 | 0

32. Secondary Outcome: Number of Participants With Any Outpatient Visits
Description: Number of participants with any outpatient visit (Health Care Professional Visit or Referral) were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 87 | 9

33. Secondary Outcome: Total Number of Outpatient Visits
Description: Total number of outpatient visit (Health Care Professional Visit or Referral) were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Number; unit: Outpatient visits
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Outpatient visits | 103 | 12

34. Secondary Outcome: Type of Outpatient Visits
Description: Type of outpatient visit (Health Care Professional Visit or Referral) such as secondary care visit (specialist), secondary care referral (specialist), primary care visit (general practitioner) and emergency room (ER) visit were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 87 | 9
Participants
  Secondary care visit (specialist) | 70 | 9
  Secondary care referral (specialist) | 15 | 1
  Primary care visit (general practitioner) | 6 | 0
  ER visit | 4 | 1

35. Secondary Outcome: Duration Between Isavuconazole Treatment Initiation and First Outpatient Visit
Description: Duration between Isavuconazole treatment was defined as the date of first outpatient visit minus the date of isavuconazole treatment initiation. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 85 | 8
Days | 63.0 (78.2) | 82.6 (128.0)

36. Secondary Outcome: Number of Participants With Inpatient Hospitalization
Description: Number of participants according to index treatment administered in the inpatient setting were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants | 114 | 14

37. Secondary Outcome: Number of Participants With Primary Reason For Inpatient Hospitalization
Description: Number of participants with primary reason for inpatient hospitalization such as other disease monitoring, other, invasive aspergillosis or mucormycosis disease monitoring, AE related to invasive aspergillosis or mucormycosis and unknown were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 114 | 14
Participants
  Other disease monitoring | 83 | 8
  Other | 31 | 6
  Invasive aspergillosis or mucormycosis disease monitoring | 27 | 2
  AE related to invasive aspergillosis or mucormycosis | 2 | 0
  Unknown | 2 | 0

38. Secondary Outcome: Duration Between Isavuconazole Treatment Initiation and Inpatient Hospitalization
Description: Duration between Isavuconazole treatment was defined as the date of inpatient hospitalization minus the date of isavuconazole treatment initiation. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 113 | 13
Days | 65.2 (108.8) | 77.2 (125.1)

39. Secondary Outcome: Mean Length of Stay For Inpatient Hospitalization
Description: Length of stay was computed as the date of discharge from hospital minus the date of hospitalization plus (+) 1. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 113 | 13
Days | 20.8 (44.3) | 20.0 (23.7)

40. Secondary Outcome: Number of Participants According to Location for Inpatient Hospitalization
Description: Number of participants according to location for inpatient hospitalization such as: hematology ward, other ward, intensive care unit, transplantation ward, emergency room, general medicine ward, oncology ward and unknown were reported in this outcome measure. Index date was defined as date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Aspergillosis | Mucormycosis
Number analyzed (Participants) | 201 | 17
Participants
  Haematology ward | 61 | 6
  Other ward | 40 | 5
  Intensive unit care (ICU) | 21 | 1
  Transplantation ward | 14 | 1
  Emergency room (ER) | 9 | 3
  General medicine ward | 9 | 0
  Oncology ward | 6 | 2
  Unknown | 2 | 0

ADVERSE EVENTS:
Time Frame: From index date until 6 months after post-index treatment discontinuation, death, or loss to follow-up, whichever occurred first (retrospective data extracted and evaluated from study start date and until study completion, approximately 34 months); Index date: date of Isavuconazole treatment initiation anytime in between 15 October 2015 until 30 June 2019
Description: Same event may appear as non-SAE and SAE, however, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Invasive Aspergillosis | Mucormycosis
All-Cause Mortality (participants affected / at risk) | 127/201 | 10/17
Serious Adverse Events (participants affected / at risk) | 34/201 | 3/17
Other Adverse Events (participants affected / at risk) | 17/201 | 2/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Invasive Aspergillosis (N=201) | Mucormycosis (N=17)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Clostridium difficile infection (Gastrointestinal disorders) | 1 | 1
Acute Gastrointestinal, Graft-versus-host disease (GVHD) (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Allergic reaction (General disorders) | 1 | 0
Multiorgan failure (General disorders) | 1 | 0
Anorexia (General disorders) | 1 | 0
Paraesthesia (General disorders) | 1 | 0
Hemoptosis (General disorders) | 1 | 0
Delerium (Nervous system disorders) | 1 | 0
Myopathy (Nervous system disorders) | 1 | 0
Intracerebral haemorrhage (Nervous system disorders) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Progression of Invasive fungal disease (Infections and infestations) | 1 | 0
Hypogammaglobulinaemia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopaenia (Blood and lymphatic system disorders) | 1 | 1
Haematological recurrence (Blood and lymphatic system disorders) | 1 | 0
Hypokalaemia (Blood and lymphatic system disorders) | 1 | 0
Hyperkalaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropaenia (Blood and lymphatic system disorders) | 1 | 1
Gamma-glutamyl transferase (Blood and lymphatic system disorders) | 1 | 0
Abnormal liver chemistry test (Blood and lymphatic system disorders) | 5 | 1
Epistaxis (Blood and lymphatic system disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Cheilitis (Skin and subcutaneous tissue disorders) | 0 | 1
Shingles (Skin and subcutaneous tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Cardio-respiratory shock (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cardio-respiratory Failure (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Stem cell transplantation (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Surgery (Surgical and medical procedures) | 1 | 1
Aspergillosis cyst removal (Surgical and medical procedures) | 1 | 0
Choreotinitis (General disorders) | 0 | 1
Castelman's disease relapse (General disorders) | 1 | 1
Renal failure (General disorders) | 1 | 1
Death (General disorders) | 15 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Invasive Aspergillosis (N=201) | Mucormycosis (N=17)
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Phlebitis (General disorders) | 0 | 1
Peripheral oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hypoacusis (Nervous system disorders) | 1 | 0
Myopathy (Nervous system disorders) | 2 | 0
Hallucinations (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Hypogammaglobulinaemia (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopaenia (Blood and lymphatic system disorders) | 1 | 0
Hypokalaemia (Blood and lymphatic system disorders) | 1 | 0
Hyperkalaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropaenia (Blood and lymphatic system disorders) | 1 | 0
Gamma-glutamyl transferase increase (Blood and lymphatic system disorders) | 1 | 0
Abnormal liver chemistry test (Blood and lymphatic system disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Cheilitis (Skin and subcutaneous tissue disorders) | 1 | 0
Shingles (Skin and subcutaneous tissue disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT04550936/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT04550936/SAP_001.pdf